CLINICAL TRIAL: NCT01322945
Title: Observational Study of Nasal Outcomes Following Endonasal Surgery for Anterior Skull Base Lesions
Brief Title: Barrow Nasal Inventory Survey
Acronym: BNI
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 10BN172
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Pituitary Tumors
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endonasal surgery: Single cohort of patients undergoing endonasal surgery

SUMMARY:
The purpose of this study is to evaluate patient nasal outcome following endo-nasal surgery. This type of surgery is conducted for pituitary and skull base tumors. There is no published data on trauma to the nose during surgery and how it impacts nasal functioning. The investigators propose to develop a survey and administer it to patients before and after surgery to learn about their perception of nasal functioning.

DETAILED DESCRIPTION:
A 9-item patient survey (the ASK Nasal Inventory) focusing on the most common postoperative complaints, such as crusting, sinusitis, pain, and ease of breathing, was developed by the anterior skull base team at the Barrow Neurological Institute. Content was validated in structured patient interviews by four subject-matter experts with both endonasal and control groups. Eligible patients for the control group included patients undergoing any neurosurgical procedure requiring anesthesia that did not involve the endonasal corridor, such as spinal decompression procedures, craniotomies for trigeminal neuralgia, and shunting procedures. This survey was self-administered pre- and 3 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults with planned endonasal surgery for pituitary tumor or skull base lesion

Exclusion Criteria:

* Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgery and endocrinology clinic
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Little, MD, Principal Investigator — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

REFERENCES:
- [Result] Little AS, Jahnke H, Nakaji P, Milligan J, Chapple K, White WL. The anterior skull base nasal inventory (ASK nasal inventory): a clinical tool for evaluating rhinological outcomes after endonasal surgery for pituitary and cranial base lesions. Pituitary. 2012 Dec;15(4):513-7. doi: 10.1007/s11102-011-0358-4. PMID 22038032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible adult patients were identified in the outpatient neurosurgical clinics at the Barrow Neurological Institute between October 2010 and June 2011.
Groups:
- Endonasal Group: Patients undergoing endonasal surgery for anterior skull base tumors, pituitary tumors, and skull base spinal fluid leaks using endonasal techniques.
- Control Group: Patients undergoing any neurosurgical procedure requiring general anesthesia that did not involve the endonasal corridor, such as spinal decompression procedures, craniotomies for trigeminal neuralgia, or shunting procedures.
Period: Overall Study
Arm/Group | Endonasal Group | Control Group
Started | 52 | 42
Completed | 52 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endonasal Group | Control Group | Total
Number analyzed (Participants) | 52 | 42 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 32 | 73
  >=65 years | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15.49) | 54.17 (14.83) | 50.27 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 27 | 18 | 45
Region of Enrollment [Number; unit: participants]
  United States | 52 | 42 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Survey Response From Baseline to 90 Days Post Surgery
Description: Mean survey response at 90 days post surgery between the control patients and the endonasal surgery patients using the Anterior skull base nasal inventory (ASK Nasal Inventory. A 5-point Likert scale for each question on the ASK Nasal inventory measures frequency of nasal symptoms where 1=never, 2= a little of the time, 3=some of the time, 4=most of the time, 5= all of the time. Total mean Likert scores were compared in the endonasal group to the control group after surgery. Scores range from minimum of 9 to maximum of 45. The lower the score the fewer the nasal complaints.
Time Frame: Baseline, 90 days post surgery
Population: Power analyses were conducted to determine a sample size large enough to significantly detect change with 90% power using a pre- post research methodology.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endonasal Group | Control Group
Number analyzed (Participants) | 52 | 42
units on a scale | 17.3 (6.7) | 13.5 (4.2)
Statistical Analysis 1: Comparison: Endonasal Group vs Control Group; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Test-retest Reliability of the ASK Nasal Inventory
Description: First 12 endonasal and 10 control patients enrolled in the study completed the ASK Nasal Inventory at 90 days and 120 days post surgery to measure reliablity of the survey (they scored the 9-item instrument similarly at both time frames)comparing 5-point Likert scale scores. Pearson correlation was used to determine a correlation between each patient's responses at 90 days post op and 120 days post op.
Time Frame: 90 days and 120 days post surgery
Measure: Number; unit: Correlation Coefficient
Groups:
- Endonasal Group: First 12 patients enrolled undergoing endonasal surgery for anterior skull base tumors, pituitary tumors, and skull base spinal fluid leaks using endonasal techniques.
- Control Group: First 10 patients enrolled undergoing any neurosurgical procedure requiring general anesthesia that did not involve the endonasal corridor, such as spinal decompression procedures, craniotomies for trigeminal neuralgia, or shunting procedures.
Arm/Group | Endonasal Group | Control Group
Number analyzed (Participants) | 12 | 10
Correlation Coefficient | 0.87 | 0.95

ADVERSE EVENTS:
Arm/Group | Endonasal Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/42
Other Adverse Events (participants affected / at risk) | 0/52 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No